CLINICAL TRIAL: NCT04765306
Title: Fascial Closure Technique After Gynecologic Laparoscopic Surgery and Postoperative Pain: a Randomized Controlled Trial
Brief Title: Fascial Closure Technique After Gynecologic Laparoscopic Surgery and Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jessica G Putman (Other)
Responsible Party: Sponsor-Investigator, Jessica G Putman, Fellow Investigator, University of Tennessee
Organization: University of Tennessee (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-004
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Masking Description: This will be a prospective, singled-blinded, randomized controlled study. Eligible patients who provide consent will be randomized into one of two arms either undergoing fascial closure with a fascial closure device or traditional direct closure on the day of surgery. Every patient will have equal probability of being assigned to either study arm. The patients will be blinded to which study arm they have been assigned to, but providers will be aware due to the nature of study topic.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Traditional Direct Fascial Closure (Active Comparator): At the beginning of the laparoscopic procedure, all patients will receive 5 mL of 0.5% ropivacaine into each laparoscopic incision site. Patients in this group will have fascia closed under traditional direct visualization without laparoscopic guidance using a single interrupted suture of 0-vicryl.
  Interventions: Device: Traditional Direct Fascial Closure
- Fascial Closure Device (Active Comparator): At the beginning of the laparoscopic procedure, all patients will receive 5 mL of 0.5% ropivacaine into each laparoscopic incision site. Patients in this group will have fascia closed using direct laparscopic visualization with the Carter-Thomason fascial closure device with a single interrupted suture of 0-vicryl.
  Interventions: Device: Fascial Closure Device

INTERVENTIONS:
Device: Traditional Direct Fascial Closure — Fascial closure using traditional surgical instruments and suture without laparoscopic guidance.
  Arms: Traditional Direct Fascial Closure
Device: Fascial Closure Device — Fascial closure using a fascial closure device under direct laparoscopic guidance.
  Arms: Fascial Closure Device

SUMMARY:
Our study aims to determine postoperative pain outcomes when comparing port site > 10 mm fascial closure with traditional direct closure versus use of laparoscopic fascial closure device in patients undergoing minimally invasive gynecologic surgery via laparoscopic or robotic techniques. Pain outcomes will be measured using the visual analog scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or older.
* Any patient undergoing laparoscopic gynecologic surgery with one left upper quadrant port site > 10 mm via either robotic or traditional laparoscopic techniques for any indication including abnormal bleeding, pelvic pain, gynecologic cancer, uterine fibroids, etc. Procedures performed will include but not be limited to hysterectomy, bilateral or unilateral salpingoophorectomy, ovarian cystectomy, and pelvic floor support procedures.
* Patients willing and able to give informed consent.
* Patients capable and willing to return for follow up and complete pain diaries.

Exclusion Criteria:

* Patients unable to return for follow up.
* Patients undergoing laparoscopic surgery that requires conversion to laparotomy.
* Patients undergoing laparoscopic surgery that does not require a port site >10 mm.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
Postoperative pain scores via Visual Analog Scale | Through 2 weeks postoperatively
  A 20 mm difference in VAS score and a 2-unit difference on a 10-point pain scale have been described as a clinically significant difference between treatment groups.

SECONDARY OUTCOMES:
Quantity of narcotics consumed in postoperative period | Through 2 weeks postoperatively
  Number of tablets of narcotics consumed in postoperative period
Length of hospital stay | Through study completion, up to 6 months
  Length of hospital stay in days from day of surgery until discharge home
Postoperative complication | Through 6 weeks postoperatively
  Postoperative incisional infection, postoperative incisional hernia
Fascial closure operating time | Duration of fascial closure operating time
  Timing of fascial closure will start when the surgeon or surgical assistant reports s/he is beginning the fascial closure and stop after the suture is cut after tying.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Boren, MD, Principal Investigator — University of Tennessee College of Medicine Gynecology Oncology; Jessica G Putman, MD, Study Director — University of Tennessee Chattanooga Minimally Invasive Gynecologic Surgery Fellow
Locations (1):
- Erlanger Baroness Hospital, Chattanooga, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No